CLINICAL TRIAL: NCT00397865
Title: A Primary Care Educational Intervention for Families of Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2006-1259
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-07

CONDITIONS: Obesity
Keywords: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: Educational booklet

INTERVENTIONS:
Behavioral: Educational booklet — Parental perception of educational booklet and evaluating any change in child's weight.

SUMMARY:
The purpose of the research is to find out if an educational booklet is helpful to families with overweight children. The educational booklet contains information for parents about nutritious eating, physical activity, and strategies for healthy living.

DETAILED DESCRIPTION:
The prevalence of overweight among children has at least doubled in the past 25 years. In the year 2004, 18.8% of children ages 6-11 were overweight. Being overweight as a child is clearly associated with adulthood obesity. In addition, complications once prevalent only in adults are now being seen in overweight children and adolescents. These include hypertension, hypercholesterolemia, and type II diabetes which are well known risk factors for cardiovascular disease. Obesity is also associated with low self-esteem among some groups of overweight adolescents.

Primary care providers are in a unique position to combat this epidemic. However, a recent survey found that only 12% of pediatricians felt highly effective in their ability to treat obesity. Furthermore, physicians reported that low self-efficacy in treating obesity was associated with a lack of patient educational materials. Few written resources for families of overweight children have been tested in the primary care setting. Much of the research on childhood overweight has been conducted in specialty obesity clinics where the resources and patient population may differ from those of primary care offices.

Kid STRIDE is an educational booklet designed for parents of overweight children. It includes information about nutrition, physical activity, and strategies for healthy living. It is hypothesized that the booklet will be distributed to and used by parents of children who are overweight or at risk for overweight. This study will analyze parents' perceptions of this booklet in order to improve its potential value. Information obtained from this pilot study will be used to prepare for a future study to determine the effectiveness of this intervention.

The purpose of this study is:

Aim 1 is to determine the distribution rate and uptake rate of an educational booklet for parents of children between the ages of 8 and 12 who are overweight.

Aim 2 is to describe parents' perceptions of the educational booklet.

Aim 3 is to assess the impact of the intervention on BMI as measured by change in BMI z-score.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to the 95th percentile for age and gender
* Presenting to pediatrician for a health maintenance visit

Exclusion Criteria:

* Genetic conditions known to predispose to overweight
* Endocrine conditions associated with overweight
* Chronic steroid therapy
* Current enrollment in a professional weight management program

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2006-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Describe parents' perceptions of the educational booklet | one year
Determine the uptake rate of an educational booklet for parents of overweight children between the ages of 7 and 12 | 6 months
Assess the impact of the intervention on BMI as measured by change in BMI z-score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - UW East Towne Pediatric Clinic, Madison, Wisconsin
  - Associated Physicians Pediatric Clinic, Madison, Wisconsin
  - Boys & Girls Club of Dane County, Madison, Wisconsin
  - UW West Pediatric Clinic, Madison, Wisconsin

REFERENCES:
- [Background] Whitlock EP, Williams SB, Gold R, Smith PR, Shipman SA. Screening and interventions for childhood overweight: a summary of evidence for the US Preventive Services Task Force. Pediatrics. 2005 Jul;116(1):e125-44. doi: 10.1542/peds.2005-0242. PMID 15995013
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Guo SS, Roche AF, Chumlea WC, Gardner JD, Siervogel RM. The predictive value of childhood body mass index values for overweight at age 35 y. Am J Clin Nutr. 1994 Apr;59(4):810-9. doi: 10.1093/ajcn/59.4.810. PMID 8147324
- [Background] Freedman DS, Dietz WH, Srinivasan SR, Berenson GS. The relation of overweight to cardiovascular risk factors among children and adolescents: the Bogalusa Heart Study. Pediatrics. 1999 Jun;103(6 Pt 1):1175-82. doi: 10.1542/peds.103.6.1175. PMID 10353925
- [Background] Strauss RS. Childhood obesity and self-esteem. Pediatrics. 2000 Jan;105(1):e15. doi: 10.1542/peds.105.1.e15. PMID 10617752
- [Background] Perrin EM, Flower KB, Garrett J, Ammerman AS. Preventing and treating obesity: pediatricians' self-efficacy, barriers, resources, and advocacy. Ambul Pediatr. 2005 May-Jun;5(3):150-6. doi: 10.1367/A04-104R.1. PMID 15913408